CLINICAL TRIAL: NCT01902030
Title: Diagnostic Study of Performance of an Aspergillus Specific Polymerase Chain Reaction in Tissue and Pleural Effusion Samples of Immunocompromised Patients for the Diagnosis of Invasive Aspergillosis
Brief Title: Evaluation of Performance of An Aspergillus PCR in Tissue and Pleural Effusion Samples of Immunocompromised Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Dieter Buchheidt, MD, Heidelberg University
Other Study IDs: ASP PCR IA TISSUE-EFFUSION
Record Dates: First submitted 2013-06-27; First posted 2013-07-17 (Estimated); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Aspergillosis; Immunosuppression
MeSH Terms: conditions — Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Fungal DNA, no human DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Proven/Probable IA Patients: Case Population
- possible/No IA Patients: Control population

SUMMARY:
Although being a frequent and lethal complication in patients (pts) with hematologic malignancies, diagnosing invasive aspergillosis (IA) still remains a difficult issue as culture-based methods show low sensitivity especially under the current clinical practice of antifungal prophylaxis or rapid antifungal therapy. In certain clinical settings, performing biopsies for identification of the underlying infectious organism becomes important. However, as culture-based methods only yield results in a minority of patients, using non-culture-based methods like Aspergillus specific polymerase chain reaction (PCR) for detection of IA directly in clinical specimens is becoming increasingly important and might help to characterize the causative pathogen.

Therefore the performance of an established Aspergillus-specific nested PCR in biopsies, re-section material or pleural effusions is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised individuals with suspicion of harbouring an invasive fungal infection
* Definition by 2008 EORTC/MSG Criteria (de Pauw CID 2008)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Immunocompromised individuals with suspicion of harbouring an invasive fungal infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Calculation of sensitivity, Specificity, positive predictive value, negative predictive value and diagnostic odds ratio | 3 months
  Evaluation of Sensitivity, Specificity, positive predictive value, negative predictive value and diagnostic odds ratio of aspergillus specific PCR in tissue and effusion samples by comparing the population with proven / probable invasive aspergillosis with patients suffering from No IA according to recent EORTC/MSG criteria of PCR in Biopsies/Effusion samples of Patients

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Buchheidt, MD, Principal Investigator — Heidelberg University
Locations (12):
- Germany (12):
  - Cologne University Hospital, Cologne
  - Duesseldorf University Hospital, Düsseldorf
  - Eschweiler General Hospital, Eschweiler
  - Frankfurt (Oder) General Hospital, Frankfurt (Oder)
  - Freiburg University Hospital, Freiburg im Breisgau
  - Halle University Hospital, Halle
  - Thoraxklinik at Heidelberg University Hospital, Heidelberg
  - Marienhospital Herne, Herne
  - Mannheim University Hospital, Mannheim
  - Prosper Hospital Recklinghausen, Recklinghausen
  - Wiesbaden Bone Marrow transplantation center, Wiesbaden
  - Wuerzburg University Hospital, Würzburg

REFERENCES:
- [Background] Spiess B, Seifarth W, Hummel M, Frank O, Fabarius A, Zheng C, Morz H, Hehlmann R, Buchheidt D. DNA microarray-based detection and identification of fungal pathogens in clinical samples from neutropenic patients. J Clin Microbiol. 2007 Nov;45(11):3743-53. doi: 10.1128/JCM.00942-07. Epub 2007 Aug 22. PMID 17715373
- [Derived] Boch T, Reinwald M, Postina P, Cornely OA, Vehreschild JJ, Heussel CP, Heinz WJ, Hoenigl M, Eigl S, Lehrnbecher T, Hahn J, Claus B, Lauten M, Egerer G, Muller MC, Will S, Merker N, Hofmann WK, Buchheidt D, Spiess B. Identification of invasive fungal diseases in immunocompromised patients by combining an Aspergillus specific PCR with a multifungal DNA-microarray from primary clinical samples. Mycoses. 2015 Dec;58(12):735-45. doi: 10.1111/myc.12424. Epub 2015 Oct 26. PMID 26497302